CLINICAL TRIAL: NCT03135301
Title: Efficacy of Combined Letrozole-metformin in Comparison With Letrozole Only in Clomiphene Resistant Infertile Women With Polycystic Ovarian Syndrome
Brief Title: Letrozole in Clomiphene Resistant Infertile Women With Polycystic Ovarian Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LET
Record Dates: First submitted 2017-04-27; First posted 2017-05-01 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Letrozole; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- letrozole plus metformin (Experimental): 5 mg of letrozole will be administered only for 5 days from day 3 each month of spontaneous or induced bleeding plus metformin will be started from the first day with a dose of 850 mg (1 tablet daily) and the dosage will be increased after 1 week up to 1,700 mg/day (2 tablets daily) and will be continued
  Interventions: Drug: letrozole plus metformin
- letrozole (Active Comparator): 5 mg of letrozole will be administered only for 5 days from day 3 each month of spontaneous or induced bleeding
  Interventions: Drug: letrozole

INTERVENTIONS:
Drug: letrozole plus metformin — letrozole 5 milligram tablets plus metformin 850 milligram tablets
  Arms: letrozole plus metformin
Drug: letrozole — letrozole 5 milligram tablets
  Arms: letrozole

SUMMARY:
Polycystic ovary syndrome accounts for the vast majority of anovulatory symptoms and hyperandrogenism in women. The diagnosis of Polycystic ovary syndrome has life-long implications, with increased risk for infertility, metabolic syndrome, and type 2 diabetes mellitus, and possibly for cardiovascular disease and endometrial carcinoma. Polycystic ovary syndrome is diagnosed in adolescents with otherwise unexplained, persistent hyperandrogenic anovulatory symptoms that are inappropriate for age and stage of adolescence. It should be considered in any adolescent girl with a chief complaint of hirsutism, treatment-resistant acne, menstrual irregularity, acanthosis nigricans, and/or obesity

ELIGIBILITY:
Inclusion Criteria:

* polycystic ovaries patients who had failed to become pregnant after 3 courses of 150 mg of clomiphene citrate (considered as clomiphene resistant),whereas the value of the above mentioned investigation are normal.

Exclusion Criteria:

1. women with other causes of infertility as male factor,tubal factor,those with endocrine disorders as thyroid dysfunction and hyperprolactinemia.
2. women who received hormonal treatment or ovulation induction drugs in the last 3 months before the study.
3. women with history of liver,kidney or cardiovascular disease.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-06-20 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
The ovulation rate | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Franik S, Le QK, Kremer JA, Kiesel L, Farquhar C. Aromatase inhibitors (letrozole) for ovulation induction in infertile women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2022 Sep 27;9(9):CD010287. doi: 10.1002/14651858.CD010287.pub4. PMID 36165742